CLINICAL TRIAL: NCT06643195
Title: Immediate Allogeneic Hematopoietic Stem Cell Transplantation Versus Re-treatment for Patients With High-Risk Acute Myeloid Leukemia: a Randomised, Open-label, Phase 2 Clinical Trial.
Brief Title: Immediate Allogeneic Hematopoietic Stem Cell Transplantation Versus Re-treatment for Patients With High-Risk Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024063
Record Dates: First submitted 2024-09-22; First posted 2024-10-16 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: AML
Keywords: High-Risk Acute Myeloid Leukemia
MeSH Terms: interventions — Retreatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disease control group (Experimental): patients proceeded to allogeneic HSCT as soon as possible. Patients were allowed to receive low-dose chemotherapy that is not intended for the purpose of achieving a second remission.
  Interventions: Other: ImmediateAllogeneic Hematopoietic Stem Cell Transplantation
- Retreatment group (Active Comparator): Receive a second course of anti-leukemic treatment prior to allogeneic HSCT. The anti-leukemic treatment regimen will be determined based on the genetic mutation status. Patients without targetable mutations will receive a combination of BCL-2 inhibitors and demethylating agents as salvage chemotherapy. Patients with targetable mutations will receive appropriate targeted therapy (e.g., FLT3 inhibitors, IDH inhibitors).
  Interventions: Other: Retreatment

INTERVENTIONS:
Other: ImmediateAllogeneic Hematopoietic Stem Cell Transplantation — patients proceeded to allogeneic HSCT as soon as possible. Patients were allowed to receive low-dose chemotherapy that is not intended for the purpose of achieving a second remission.
  Arms: Disease control group
Other: Retreatment — Receive a second course of anti-leukemic treatment prior to allogeneic HSCT. The anti-leukemic treatment regimen will be determined based on the genetic mutation status. Patients without targetable mutations will receive a combination of BCL-2 inhibitors and demethylating agents as salvage chemotherapy. Patients with targetable mutations will receive appropriate targeted therapy (e.g., FLT3 inhibitors, IDH inhibitors).
  Arms: Retreatment group

SUMMARY:
This study aims to investigate whether immediate HSCT for patients with high-risk AML and intermediate-risk AML who have not achieved complete remission (CR) after their first induction therapy is non-inferior to re-treatment with chemotherapy.

DETAILED DESCRIPTION:
1. Disease control group: patients proceeded to allogeneic HSCT as soon as possible. Patients were allowed to receive low-dose chemotherapy that is not intended for the purpose of achieving a second remission.
2. Retreatment group: Receive a second course of anti-leukemic treatment prior to allogeneic HSCT. The anti-leukemic treatment regimen will be determined based on the genetic mutation status. Patients without targetable mutations will receive a combination of BCL-2 inhibitors and demethylating agents as salvage chemotherapy. Patients with targetable mutations will receive appropriate targeted therapy (e.g., FLT3 inhibitors, IDH inhibitors).

For patients who have already received targeted therapy during induction treatment, the researchers may choose the treatment regimen based on the individual patient's condition.

ELIGIBILITY:
Inclusion Criteria:

1. AML patients aged ≥ 18 years.
2. High-risk AML patients according to the 2022 ELN standards who received one cycle of induction therapy.
3. Requires allogeneic hematopoietic stem cell transplantation (including HLA-matched or mismatched allogeneic HSCT and unrelated donor transplant).
4. KPS score greater than 60.
5. Informed consent must be signed before the start of the study procedures; if it is detrimental to the patient's condition for them to sign, the consent may be signed by a legal guardian or immediate family member.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Patient has received more than 440 mg/m2 daunorubicin equivalents. The cumulative dose is calculated by summing up isotoxic daunorubicin-equivalents for daunorubicin, doxorubicin, epirubicin, idarubicin and mitoxantrone. The conversion factors are derived from the comparison of the respective maximum doses. The conversion factor is 1 for daunorubicin, 1 for doxorubicin, 0.6 for epirubicin, 4.6 for idarubicin, and 2.7 for mitoxantrone (see worksheet for calculation).
3. Severe organ dysfunction, defined as:

1) Left ventricular ejection fraction <50%. 2) Patients who receive supplementary continuous oxygen. 3) Serum bilirubin >1.5 x ULN (if not considered Gilbert-Syndrome) or ASAT/ALAT >5 x ULN.

4) Estimated Glomerular Filtration Rate (GFR) < 50 ml/min, where: Estimated GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.203 x (0.742 if patient is female) x (1.212 if patient is black) 4. History of allogeneic transplantation. 5. Manifestation of AML in the Central Nervous System. 6. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
treatment success | day 56 after allogeneic HCT
  The primary endpoint, treatment success defined as complete remission on day 56 after allogeneic HCT, was defined as dichotomous success rate.

SECONDARY OUTCOMES:
Cumulative Incidences of Allogeneic HSCT | HSCT rates at 4,8,16, and 24 weeks
  1. Starting point: Randomization
  2. Event: allogeneic HCT
  3. Competing events: death, withdrawal
Incidence of Complete Remission from Randomisation | Date of first documented CR or CRi or CRchim Death before CR/CRi/CRchim not achieve a CR or CRi by six months
  1. Starting point: randomization
  2. Event: Date of first documented CR or CRi or CRchim
  3. Competing Event: Death before CR/CRi/CRchim
  4. Administrative Censoring: not achieve a CR or CRi by six months
  b) Starting point: day 56 c) Events: Relapse (both, hematologic or molecular) and death
Overall survival after HCT | Death
  1. Starting point: HCT
  2. Event: Death
Event-free survival after HCT | death before relapse, relapse (both, hematological or molecular), and failure to achieve a CR at final remission assessment
  1. Starting point: HCT
  2. Events: death before relapse, relapse (both, hematological or molecular), and failure to achieve a CR at final remission assessment
Leukemia-free survival from day 56 after alloHCT for patients who met the primary endpoint | day 56
  efined only for per-protocol treated patients who met the primary endpoint b) Starting point: day 56 c) Events: Relapse (both, hematologic or molecular) and death
Rate of MRD Negative from Day 56 after HSCT | day 56
  1. defined only for per-protocol treated patients who met the primary endpoint
  2. Starting point: day 56
  3. Events: MRD Negative (including MPFC, qPCR and NGS) and death
7. Overall Survival from Randomization: Measured from the start of randomization, with the primary event being death. | Death
  1. Starting point: Randomization
  2. Event: Death

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hebei Medical University Second Hospital, Shijiazhuang, Hebeisheng
  - Zhengzhou University First Affiliated Hospital, Zhengzhou, Henan
  - The 960th Hospital of the Joint Service Support Force of the Chinese People's Liberation Army, Jinan, Shandong
  - People's Liberation Army The General Hospital of Western Theater Command, Chengdu, Sichuan